CLINICAL TRIAL: NCT01101906
Title: A Randomized, Placebo-controlled, Double-blinded Phase 2 Study of Second-line Treatment With OSI-906 in Patients With Advanced Hepatocellular Carcinoma (HCC) After Failure of First-line Treatment With Sorafenib
Brief Title: A Randomized, Placebo-controlled, Double-blind Phase 2 Study With OSI-906 in Patients With Advanced HCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decided not to pursue the development of this drug in this patient population at this time
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OSI-906-206; 2010-018739-17 (EudraCT Number)
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
Keywords: HCC; OSI-906; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: OSI-906 (Experimental): 150 mg BID
  Interventions: Drug: OSI-906
- Arm B: Placebo (Placebo Comparator): Placebo BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OSI-906 — OSI-906 administered orally
  Arms: Arm A: OSI-906
Drug: Placebo — Matching placebo administered orally
  Arms: Arm B: Placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blind phase 2 study of OSI-906 or placebo at a continuous 150 mg twice daily (BID) dose.

DETAILED DESCRIPTION:
Adult patients with advanced HCC previously treated with sorafenib will be randomized 2:1 to receive either single agent OSI-906 or placebo

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of advanced HCC. Clinical diagnosis by American Association for the Study of Liver Diseases (AASLD) criteria in cirrhotic patients is acceptable. For patients without cirrhosis histological confirmation is mandatory
* Patients must have received prior systemic treatment for advanced HCC with sorafenib and had confirmed disease progression or had discontinued sorafenib due to a drug related toxicity
* Patient has received their last dose of sorafenib at least 14 days prior to randomization
* Patient has recovered from sorafenib or investigational agent related toxicity to ≤ grade 2
* Measurable disease according to RECIST (version 1.1)
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 - 1
* Child-Pugh Status A or B(7)
* Barcelona Clinic Liver Cancer (BCLC) stage B/C
* Previous local therapy (eg, surgery, radiation therapy, hepatic arterial therapy, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation) is permitted if ≥ 21 days before randomization
* Fasting glucose ≤ 150 mg/dL (8.3 mmol/L). Concurrent use of non-insulinotropic oral antihyperglycemic therapy is permitted if the dose has been stable for ≥ 4 weeks at the time of randomization
* Following laboratory parameters (determined by laboratory):

  * Platelets ≥ 60 x 10^9/L
  * Hemoglobin ≥ 8.5 g/dL
  * Absolute neutraphil count (ANC) ≥ 1.5 x 10^9/L
  * Potassium within normal limits (supplementation may be used)
  * Partial thrombopastin time (PTT) ≤ 2.3 x Upper Limit of Normal (ULN)
  * Magnesium within normal limits (supplementation may be used)
  * Calcium within normal limits (supplementation may be used)
* Adequate organ function (for a HCC population):

  * Liver function test (LFT) ≤ 5 x ULN
  * Albumin ≥ 2.8 g/dL
  * Total bilirubin ≤ 2.8 mg/dL
  * Creatinine ≤ 1.5 x ULN
  * International normalized ratio (INR) ≤ 2.3
* Estimated life expectancy ≥ 12 weeks based on an investigator assessment of recent changes in laboratory values, performance status, and other clinical criteria
* Patients, both males and females, with reproductive potential (ie, menopausal for less than 1 year and not surgically sterilized) must agree to practice effective contraceptive measures throughout the study. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to randomization
* Patients must provide written informed consent to participate in the study
* Prior radiation therapy is permitted provided patients have recovered from the acute, toxic effects of radiotherapy prior to randomization. A minimum of 21 days must have elapsed between the end of radiotherapy and randomization; and
* Prior surgery is permitted provided that the surgery was done ≤ 28 days prior to randomization and adequate wound healing has occurred prior to randomization

Exclusion Criteria:

* Child-Pugh B (8 - 9) or C
* Patients who are candidates for potentially curative intervention (ie, surgical resection or transplantation)
* Type 1 diabetes mellitus or Type 2 diabetes mellitus currently requiring insulinotropic or insulin therapy
* Prior insulin-like growth factor - 1 receptor (IGF-1R) therapy
* Patients requiring interferon
* Patients with uncontrolled symptomatic ascites
* Prior investigational agent within 21 days prior to randomization
* History of poorly controlled gastrointestinal disorders that could affect the absorption of study drug (eg, Crohn's disease, ulcerative colitis, etc)
* History of organ allograft including liver transplant
* Malignancy other than HCC within the past 3 years:

  * Exceptions: resected basal cell or squamous cell carcinoma of the skin, cured in situ cervical carcinoma, cured ductal carcinoma in situ of the breast, and/or cured superficial bladder cancer
* History (within last 6 months) of significant cardiovascular disease unless the disease is well-controlled. Significant cardiac disease includes second/third degree heart block; clinically significant ischemic heart disease; superior vena cava (SVC) syndrome; poorly controlled hypertension; congestive heart failure of New York Heart Association (NYHA) Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea)
* History of arrhythmia (multifocal premature ventricular contractions [PVCs], bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) that is symptomatic or requires treatment (≥ grade 3), left bundle branch block (LBBB), or asymptomatic sustained ventricular tachycardia are not allowed. Patients with atrial fibrillation controlled by medication are not excluded
* QTcF interval at screening ≥ 450 msec
* Use of drugs that have a known risk of causing Torsades de Pointes (TdP) ('Torsades List' on www.azcert.org/medical-pros/drug-lists/by category.cfm)are prohibited within 14 days prior to randomization
* Use of the potent CYP1A2 inhibitors ciprofloxacin and fluvoxamine. Other less potent CYP1A2 inhibitors/inducers are not excluded
* History of cerebrovascular accident (CVA) within 6 months prior to randomization or that resulted in ongoing neurologic instability
* Active infection or serious underlying medical condition (including any type of active seizure disorder within 12 months prior to randomization) that would impair the ability of the patient to receive study drug
* History of human immunodeficiency virus (HIV) infection or acquired immune deficiency syndrome (AIDS)-related illness or serious acute or chronic illness
* History of any psychiatric or neurologic condition that might impair the patient's ability to understand or to comply with the requirements of the study or to provide informed consent
* Pregnant or breast-feeding females
* Symptomatic brain metastases that are not stable, require steroids, are potentially life threatening, or that have required radiation within 28 days prior to randomization; and/or
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-01-10 (Actual); Primary Completion 2011-11-04 (Actual); Study Completion 2011-12-28 (Actual)

PRIMARY OUTCOMES:
Time to progression (TTP) | 20 months
  Time from randomization to radiological disease progression based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Overall Survival (OS) | 23 months
  Date of randomization until the documented date of death
Progression Free Survival (PFS) | 23 months
  Time from randomization to radiological disease progression based on RECIST version 1.1 assessed by investigator or death due to any cause whichever occurs first
Time to Progression (including clinical progression) (TTPc) | 23 months
  Time from randomization to progression (either radiological disease progression based on RECIST version 1.1 or symptomatic clinical progression as assessed by investigator)
Disease Control Rate (DCR) | 23 months
  Proportion of patients with a best overall response of complete response (CR), partial response (PR), or stable disease based on RECIST version 1.1 criteria
Overall Response Rate | 23 months
  Proportion of patients with a best overall response of CR or PR based on RECIST version 1.1 criteria
Time to progression in patients with hepatitis B virus (HBV) and/or hepatitis C virus (HVC) | 23 months
Progression Free Survival in patients with HBV and/or HCV | 23 months
Overall Survival in patients with HBV and/or HCV | 23 months
Overall Response Rate in patients with HBV and/or HCV | 23 months
Safety assessed via physical examination, vital signs, clinical laboratory tests, electrocardiograms (ECGs) and recording adverse events | 23 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (41):
- United States (6):
  - University of California - Los Angeles, Los Angeles, California
  - Tulane University Health Services Center, New Orleans, Louisiana
  - Oregon Health & Science University, Portland, Oregon
  - Virginia Mason Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussells
  - Universitair Ziekenhuis Gent, Ghent
- France (7):
  - Hopital Jean Verdier - Dervice d'Hepato-Gastroenterologie, Bondy
  - Hôpital Henri Mondor, Créteil
  - Hopital de la Timone, Marseille
  - Hopital l'Archet 2, Nice
  - Hôpital Saint-Antoine, Paris
  - Hôpital de Tenon, Paris
  - Centre Rene Gauducheau, Saint-Herblain
- Germany (4):
  - Universitatsklinikum Essen, Essen
  - Universitätsklinikum Halle, Halle
  - Universitatsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Magdeburg A.ö.R., Magdeburg
- Queen Mary Hospital, Hong Kong, Hong Kong
- Italy (4):
  - Fondazione Ca' Granda Ospedale Maggiore Policlinico, Divisione di Gastroenterologia I, Milan
  - Ospedale Fatebenefratelli, Dipartimento Medicina Interna, Napoli
  - IRCCS Istituto Nazionale per lo studio e la cura dei tumori Fondazione G. Pascale-SSD Epatobiliare, Napoli
  - Istituto Mediterraneo per i Trapianti e Terapie ad Alta Specializzazione ISMETT-Dipartimento di Epatologia e Gastroenterologia, Palermo
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Johns Hopkins Singapore International Medical Centre, Singapore
- South Korea (6):
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela, Coruna
  - Hospital Clinic Provincial, Barcelona
  - Hospital Puerta de Hierro Majadahonda, Madrid
  - Clinica Universitaria de Navarra, Pamplona
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Chang Gung Medical Foundation LinKou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=228